CLINICAL TRIAL: NCT02816255
Title: The Efficacy of a New Mathematical Formula to Predict Continuous Positive Air Pressure With an Oronasal Mask Interface.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to budget and staff changes due to covid-19.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1602017026
Record Dates: First submitted 2016-06-23; First posted 2016-06-28 (Estimated); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-08

CONDITIONS: Obstructive Sleep Apnea (OSA)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Subjects will complete two week baseline with nasal mask then will complete two week treatment with full face either with new algorithm or old algorithm.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Full Face Mask with same CPAP Pressure (Placebo Comparator): After the two week period all will switch to a full face mask with half using the same CPAP pressure.
  Interventions: Device: Full Face Mask with same CPAP Pressure
- Full Face Mask with new Pressure (Active Comparator): After the two week period all will switch to a full face mask with half using with a new cpap pressure derived from our formula.
  Interventions: Device: Full Face Mask with new Pressure

INTERVENTIONS:
Device: Full Face Mask with same CPAP Pressure — Full Face Mask with same CPAP Pressure
  Arms: Full Face Mask with same CPAP Pressure
Device: Full Face Mask with new Pressure — New cpap pressure derived from our formula for the final two weeks.
  Arms: Full Face Mask with new Pressure

SUMMARY:
Subjects will all have a two week baseline period in which they will use a nasal mask using an air view CPAP machine (which records all data). After the two week period all will switch to a full face mask with half using the same CPAP pressure and half with a new a CPAP pressure derived from our formula for the final two weeks.

DETAILED DESCRIPTION:
The goal of this study is to test the efficacy of an algorithm the investigators previously created to adjust Continuous positive airway pressure (CPAP) when a mask interface is switched from a nasal to a full face.

Subjects will currently have a moderate to severe Apnea-hypopnea index (AHI - The Apnea-Hypopnea Index or Apnoea-Hypopnoea Index (AHI) is an index used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep). (above 15)

* Scoring of apneas Score a respiratory event as an apnea when BOTH of the following criteria are met: N1, N2, N3, N4

  1. There is a drop in the peak signal excursion by ≥90% of pre-event baseline using an oronasal thermal sensor (diagnostic study), PAP device flow (titration study) or an alternative apnea sensor (diagnostic study)
  2. The duration of the ≥90% drop in sensor signal is ≥ 10 seconds. Score an apnea as obstructive if it meets apnea criteria and is associated with absent inspiratory effort throughout the entire period of absent airflow.

     Score an apnea as central if it meets apnea criteria and is associated with absent inspiratory effort throughout the entire period of absent airflow.

     Score an apnea as mixed if it meets apnea criteria and is associated with absent inspiratory effort in the initial portion of the event, followed by resumption of inspiratory effort in the second portion of the event. N4 Note 1 - Identification of an apnea does not require a minimum desaturation criterion.

     Note 2 - If a portion of a respiratory event that would otherwise meet criteria for a hypopnea meets criteria for apnea, the entire event should be scored an apnea.

     Note 3 - If the apnea or hypopnea event begins or ends during an epoch that is scored as sleep, then the corresponding respiratory event can be scored and included in the computation of the apnea hypopnea index (AHI). This situation usually occurs when an individual; has a high AHI with events occurring so frequently that sleep is severely disrupted and epochs may end up being scored as wake even though <15 seconds of sleep is present during the epoch containing that portion of the respiratory event. However if the apnea or hypopnea occurs entirely during an epoch scored as wake, it should not be scored or counted towards the apnea hypopnea index because of the difficultly of defining a denominator in this situation. If these occurrences are a prominent feature of the polysomnogram and/or interfere with sleep onset, their presence should be mentioned in the narrative summary if the study.

     Note 4 - For alternative apnea sensors see tech specifications for Adults. There is not sufficient evidence to support a specific durations of the central and obstructive components of a mixed apnea thus specific durations of these components are not recommended.
* AASM 2015 PROTOCOL Scoring of Hypopneas Score a respiratory event as a hypopnea if all of the following criteria are met. N1, N2, N3.

  1. The peak signal excursions drop by ≥30% of pre-event baseline using nasal pressure (diagnostic study), PAP device flow (titration study), or an alternative hypopnea sensor (diagnostic study).
  2. The duration of the ≥30% drop in signal excursion is ≥10 seconds.
  3. There is a ≥3% oxygen desaturation from pre-event baseline or the event is associated with an arousal.

Subjects once consented and entered into the study, will all have a two week baseline period in which they will use a nasal mask using an airview cpap machine (which records all data). After the two week period all will switch to a full face mask with half using the same CPAP pressure and half with a new cpap pressure derived from our formula for the final two weeks.

Those placed in the randomized into a new pressure will have an experimental procedure of getting a new pressure.

The investigators expect the AHI of the controls to increase. Our two new formulas are referred to as Opred (oronasal) (full face mask) and Npred (nasal) (non-full face mask).

Npred=(0.017 AHI)-(0.092 LSaO2)+(0.225 NC)+5.534 Opred=(0.03 AHI)-(0.130 LSaO2)+19.732 NC=Neck circumference, AHI= baseline AHI, LSaO2= Lowest blood oxygen saturation from the baseline polysomnogram.

These models were developed using multiple linear regressing modeling. The study is self-funded because it has no funding. Subjects will not be compensated

ELIGIBILITY:
Inclusion Criteria:

* AHI above 15.
* Willing to switch to full face mask post titration.
* Not currently on a weight loss plan and no intention of beginning a weight loss regimen during the duration of the study

Exclusion Criteria:

* AHI below 15.
* Not willing to switch to full face mask post titration.
* Currently on a weight loss plan and / or intention of beginning a weight loss regimen during the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ebben, Ph. D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine Center for Sleep Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Full Face Mask With Same CPAP Pressure | Full Face Mask With New Pressure
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Full Face Mask With Same CPAP Pressure | Full Face Mask With New Pressure | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 4 | 4 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Severity of Sleep Apnea as Measured by the AHI
Description: The investigators will compare the Apnoea-Hypopnoea Index (AHI) of subjects with the new formula in place vs. those that don't have the formula. The Apnea-Hypopnea Index is an index used to indicate the severity of sleep apnea. It is represented by the number of apnea and hypopnea events per hour of sleep. A respiratory event is scored as an apnea when both of the following criteria are met: N1, N2, N3, N4. a) There is a drop in the peak signal excursion by greater than or equal to 90% of pre-event baseline using an oronasal thermal sensor (diagnostic study), PAP device flow (titration study) or an alternative apnea sensor (diagnostic study) b) The duration of the greater than or equal to 90% drop in sensor signal is greater than or equal to 10 seconds.
Time Frame: After a 2-week baseline period (for weeks 3 & 4), subjects will be switched from a nasal to full-face CPAP mask interface for two-weeks with either the same CPAP setting (control) or a new formula determined pressure (treatment).
Measure: Mean (Standard Deviation); unit: AHI
Arm/Group | Full Face Mask With Same CPAP Pressure | Full Face Mask With New Pressure
Number analyzed (Participants) | 6 | 5
AHI | 2.81 (1.59) | 1.59 (1.47)

2. Secondary Outcome: Lowest Oxyhemoglobin Saturation
Description: The investigators will compare the lowest oxyhemoglobin saturation of subjects with the new formula in place vs. those that don't have the formula.
Time Frame: One month
Population: We were unable to collect oximetry data in either the treatment or control groups.
Arm/Group | Full Face Mask With New Pressure | Full Face Mask With Same CPAP Pressure
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the study period which was 1-month total.
Arm/Group | Full Face Mask With New Pressure | Full Face Mask With Same CPAP Pressure
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/55/NCT02816255/Prot_SAP_000.pdf